CLINICAL TRIAL: NCT04553380
Title: Study on the Feasibility and Treatment Experience of Community Doctors in Shenzhen Guided by Specialists to Use Basic Insulin in the Treatment of Adult Type 2 Diabetes Mellitus
Brief Title: Study on the Feasibility of Community Doctors Guided by Specialists to Use Basic Insulin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YANDEWEN
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; basic insulin; community doctors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- community patient group (Experimental): The community doctor adjusts the basic insulin dosage daily according to the fasting blood glucose of the patient under the guidance of the specialist.
  Interventions: Drug: basic insulin
- inpatient group (Active Comparator): Endocrinologists in the in-patient department use the same basic insulin dose adjustment regimen to treat patients.
  Interventions: Drug: basic insulin

INTERVENTIONS:
Drug: basic insulin — 1. Initial dose of basic insulin: 0.2U/kg/d.
  2. Dose titration regimens: the dose is titrated by increments of 0.07U/kg daily until the fasting blood glucose（FBG）≤7 mmol / L, and if the FBG≤ 3.9mmol/L, the 0.07U/kg is reduced.
  3. Injection time: subcutaneous injection before going to bed every night.
  Other Names: Glargine 300U/3ml

SUMMARY:
At present, one of the reasons for the low blood sugar control rate in China is related to the late use of basic insulin and insufficient dose adjustment. If the community hospital can actively treat the diabetic patients who need to use insulin and adjust the dose in time, it will certainly improve the blood sugar control rate. However, at present, community doctors basically do not take the initiative to start insulin treatment, but only passively use insulin that has been prescribed by specialists, and there is a lack of ability to adjust the dose of insulin and treatment inertia. Therefore, it is very necessary for community doctors to receive guidance from endocrine specialists to improve their ability to use insulin. This study intends to carry out a study of endocrine specialists guiding community doctors to use basic insulin in the treatment of adult type 2 diabetes in Shenzhen Community Hospital. Through this study to understand whether the effectiveness and safety of community doctors actively using basic insulin therapy under the guidance of specialists can reach the level of specialists.

DETAILED DESCRIPTION:
The study consists of two parts: the screening period and the treatment follow-up period.

1. Screening period (day 0): patients were screened according to the inclusion and exclusion criteria, and informed consent was completed.
2. Treatment follow-up period (day 1-day 90)： Day 1： （1）all patients in the group received diet and exercise education；（2）Collect patients' basic data (name, sex, age, height, weight, waist circumference, hip circumference, etc.), detect plasma FBG and HbA1c (sent to the central laboratory for testing)；（3）Initial treatment： On the basis of the original oral medicine, the patient will initial basic insulin. The initial dose of basic insulin is 0.2U/kg/d.

Day 2-Day 89:

1. Community patient group：The community doctor adjusts the dosage of insulin daily according to the patient's FBG: the dose is titrated by increments of 0.07U/kg daily until the fasting blood glucose （FBG）≤7 mmol / L, and if the FBG≤ 3.9mmol/L, the 0.07U/kg is reduced. Inpatient group：Endocrinologists in the in-patient department use the same basic insulin dose adjustment regimen to treat patients.
2. It can be discontinued when the basic insulin is reduced to 8U and the fasting blood glucose reaches the standard for 3 days.

Day 90：Patients were re-examined the plasma FBG and HbA1c (sent to the central laboratory for testing), and community doctors filled in the treatment experience questionnaire.

Follow-up requirements: Patients use the complimentary blood glucose meter to monitor FPG every day, 2 hours postprandial blood glucose and night blood glucose are optional, and blood sugar is measured at any time if there are symptoms of hypoglycemia. The community doctor adjusted the insulin dose according to the blood glucose level every day, and the patients were followed up by telephone every week to collect the use of hypoglycemia, diet, exercise and other hypoglycemic drugs, and record the time when the FPG reached the standard, the total amount of insulin glargine, hypoglycemia and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T2DM (WHO1999 diabetes diagnostic criteria)；
2. The age is ≥ 18 and ≤ 65 years old;
3. Continuous use of 2 or more oral hypoglycemic drugs for 1 month but HbA1c ≥ 8.0% and FPG ≥ 10mmol/L.

Exclusion Criteria:

1. Severe abnormal liver and kidney function and cardiac insufficiency;
2. Complicated with all kinds of acute and chronic infection or coronary heart disease, kidney disease, connective tissue disease, tumor, stroke and so on;
3. There are acute metabolic disorders caused by stress and diseases affecting glucose metabolism, such as pheochromocytoma, acromegaly, Cushing syndrome, hyperthyroidism and so on.
4. Acute complications of diabetes, such as diabetic ketoacidosis, hyperglycemic hyperosmotic coma or lactic acidosis, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to achieve target FBG | From the beginning of intervention to fasting blood glucose ≤ 7.0mmol/L，assessed up to 3 months.
  Treatment days when FBG reached the standard (≤ 7.0mmol/L) after treatment with basal insulin.
Decrease of HbA1c | At the end of 3 months of follow-up.
  The change of HbA1c before and after treatment with basal insulin.
Incidence of hypoglycemia | At the end of 3 months of follow-up.
  The proportion of the occurrence of hypoglycemia to the number of total blood glucose monitoring.

SECONDARY OUTCOMES:
Daily doses of insulin at the study end point. | At the end of 3 months of follow-up.
  The daily doses of insulin at the study end point.

CONTACTS AND LOCATIONS:
Overall Officials: Dewen Yan, Study Chair — Shenzhen Second People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Ji L, Zhang P, Weng J, Lu J, Guo X, Jia W, Yang W, Zou D, Zhou Z, Pan C, Gao Y, Li X, Zhu D, Li Y, Wu Y, Garg SK. Observational Registry of Basal Insulin Treatment (ORBIT) in Patients with Type 2 Diabetes Uncontrolled by Oral Hypoglycemic Agents in China--Study Design and Baseline Characteristics. Diabetes Technol Ther. 2015 Oct;17(10):735-44. doi: 10.1089/dia.2015.0054. Epub 2015 Jul 14. PMID 26171728
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S98-S110. doi: 10.2337/dc20-S009. PMID 31862752
- [Background] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, DeFronzo RA, Einhorn D, Fonseca VA, Garber JR, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2019 EXECUTIVE SUMMARY. Endocr Pract. 2019 Jan;25(1):69-100. doi: 10.4158/CS-2018-0535. No abstract available. PMID 30742570